CLINICAL TRIAL: NCT00481169
Title: A Multicenter, Double Blind, Randomized, Placebo and Raloxifene Controlled Study to Assess Safety and Efficacy of TSE-424 (Bazedoxifene Acetate) in the Prevention of Postmenopausal Osteoporosis
Brief Title: Study Evaluating TSE-424/Placebo/Raloxifene in Preventing Osteoporosis in Postmenopausal Women
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 3068A1-300
Record Dates: First submitted 2007-05-30; First posted 2007-06-01 (Estimated); Last update posted 2009-08-21 (Estimated); Status verified 2009-08

CONDITIONS: Osteoporosis
Keywords: Postmenopausal Osteoporosis
MeSH Terms: conditions — Osteoporosis; Osteoporosis, Postmenopausal | interventions — bazedoxifene

INTERVENTIONS:
Drug: Bazedoxifene Acetate (TSE-424)

SUMMARY:
The purpose of this study is to determine whether TSE-424 (bazedoxifene acetate), an investigational drug, is safe and effective in the prevention of osteoporosis in postmenopausal women.

DETAILED DESCRIPTION:
Primary objective: To evaluate the safety and efficacy of 3 doses of TSE-424 (bazedoxifene acetate), an investigational drug, in comparison with those of placebo and raloxifene in preventing osteoporosis in postmenopausal women.

Secondary objective: To evaluate the effect of TSE-424 (bazedoxifene acetate), an investigational drug, in comparison with that of placebo and raloxifene on endometrium, metabolic parameters, vasomotor symptoms, adverse events, and quality of life. Samples will be collected for population pharmacokinetic (PK) analysis.

ELIGIBILITY:
Inclusion Criteria:

* Generally healthy women 45 years of age or older who are at least 1 year postmenopausal.
* Subjects must qualify for one of the following categories (a or b): a) Greater than 1 year but less than 5 years postmenopausal with at least one of the osteoporosis risk factors. b) Greater than 5 years postmenopausal with BMD T-score at lumbar spine or femoral neck between -1 and -2.5 (inclusive) with at least one osteoporosis risk factor.

Exclusion Criteria:

* One (1) or more osteoporotic vertebral fractures (T4-L4).
* Diseases that may affect bone metabolism.
* Past history or active nontraumatic venous thromboembolic events, including deep vein thrombosis, pulmonary embolism, and retinal vein thrombosis.

Min Age: 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1742 (Actual)
Dates: Start 2001-07; Primary Completion 2004-07 (Actual); Study Completion 2004-09 (Actual)

PRIMARY OUTCOMES:
The percent change from baseline in lumbar spine bone mineral density (BMD) after 24 months. | 24 months

SECONDARY OUTCOMES:
Additional BMD evaluation including total hip, femoral neck and trochanter at months 6, 12, 18 and 24. Serum bone markers at months 3, 6, 9, 12, 18 and 24. Lipid panel at months 3, 6, 12, 18 and 24. | Up to 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer